CLINICAL TRIAL: NCT01313039
Title: Evaluation of the Use of AZD6244 to Induce Increased ER Expression and Anti-Estrogen Response in ER-Negative/Low Breast Cancer
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20100252
Record Dates: First submitted 2011-03-09; First posted 2011-03-11 (Estimated); Results first posted 2014-07-02 (Estimated); Last update posted 2017-02-07 (Estimated); Status verified 2016-12

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; ER-negative; Allred Score
MeSH Terms: conditions — Breast Neoplasms | interventions — AZD 6244

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- AZD6244 (Experimental)
  Interventions: Drug: AZ6244

INTERVENTIONS:
Drug: AZ6244 — AZD6244 75 mg (3 x 25mg capsules) orally twice per day on Days 1 - 15
  Other Names: AZD6244

SUMMARY:
If AZD6244 is able to increase ER expression in ER-negative/low cancers then it may be possible to effectively use hormonal therapy in these patients resulting in improved outcomes. The investigators propose a single-arm Simon two-step study to examine whether treatment with AZD6244 will result in increased ER expression in ER-negative/low primary breast tumors.

ELIGIBILITY:
Inclusion Criteria:

* Female breast cancer patient > 18 years.
* Patients must have biopsy-proven clinical Stage Ic-III invasive breast carcinoma with ≤ 10% ER expression by immunohistochemistry (IHC) analysis.
* Patients must have a pre-treatment baseline core biopsy or incisional biopsy available for additional testing (ER, protein/gene expression analysis).
* Patients must have sufficient tumor remaining following diagnostic biopsy that requires an additional definitive surgical procedure per the standard of care. Planned procedure may include lumpectomy or mastectomy as clinically indicated.
* Patients must have an ECOG Performance Status of 0 - 1.
* Patients must have the ability to understand and willingness to sign an English or a Spanish language written informed consent document.

Exclusion Criteria:

* Male breast cancer patient.
* Patients who are pregnant or breast-feeding are excluded from the study due to potential harm to the fetus or nursing infant from the study therapy. Patients of reproductive potential must consent to use of contraception or abstinence to be eligible for the study.
* Patients may not have received prior chemotherapy or hormonal therapy for treatment of the current breast cancer.
* Patients should not have known or strongly suspected BRCA mutation by history (genetic testing not required).
* Patients will have pre-study testing, including history and physical exam, complete blood count, and measurement of renal and hepatic function. Patients will be ineligible for the study if significant abnormalities are detected, in accordance with good medical practice.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2011-02; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Judith Hurley, MD, Study Chair — University of Miami Sylvester Comprehensive Cancer Center
Locations (1):
- University of Miami Sylvester Comprehensive Cancer Center, Miami, Florida, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Single Arm: AZ6244: AZD6244 75 mg (3 x 25mg capsules) orally twice per day on Days 1 - 15
Period: Overall Study
Arm/Group | Single Arm
Started | 4
Completed | 2
Not Completed | 2
Not completed — Physician Decision | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | AZD6244
Number analyzed (Participants) | 4
Age, Continuous [Mean (Full Range); unit: years] | 59.75 [56 to 70]
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 1
Gender [Count of Participants; unit: Participants]
  Female | 4
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 4

OUTCOME MEASURES:

1. Primary Outcome: Increase of ER Protein Expression in ER-Negative/Low Breast Cancer
Description: To evaluate in a clinical neoadjuvant model whether MEK inhibitor AZD6244 can increase ER protein expression in ER-negative/low breast cancer, as measured by the "ER response rate" by both standard immunohistochemistry and Allred Score.
Time Frame: 2 years
Population: Only 1 subject had evaluable study data
Measure: Number; unit: participants
Arm/Group | Single Arm
Number analyzed (Participants) | 1
participants | 1

2. Secondary Outcome: Changes in ER-regulated Gene Expression in E-negative/Low Breast Cancer
Description: To assess for changes in ER-regulated gene expression in ER-negative/low breast tumors following AZD6244 therapy through assessment of protein expression by immunhistochemistry in paraffin embedded tissues.
Time Frame: 2 Years
Reporting Status: Not Posted

3. Secondary Outcome: Rate of ER Promoter Methylation in ER-negative/Low Breast Cancer
Description: To determine the rate of ER promoter methylation in ER-negative/low breast cancer tumors that do not attain an ER response following AZD6244 therapy.
Time Frame: 2 years
Reporting Status: Not Posted

4. Secondary Outcome: In Vitro Tamoxifen Response in Tumors
Description: To assess for in vitro tamoxifen response in tumors following therapy with AZD6244.
Time Frame: 2 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Study results not evaluated due to low accrual.
Arm/Group | Single Arm
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 0/4

LIMITATIONS AND CAVEATS:
Only 4 patients were enrolled and of these 4 only 1 patient had evaluable study data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes